CLINICAL TRIAL: NCT05328245
Title: The Effectiveness of Internet-delivered Exposure-based Cognitive Behavior Therapy for Irritable Bowel Syndrome - a Cohort Study
Brief Title: Internet-delivered Exposure-based Cognitive Behavior Therapy for Irritable Bowel Syndrome - a Cohort Effectiveness Study
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Brjann Ljotsson, Principal Investigator, Associate Professor, Karolinska Institutet
Other Study IDs: IPSY-IBS
Record Dates: First submitted 2022-03-28; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Effectiveness; Cognitive Behavioral Therapy; Exposure; Internet; Mediation
MeSH Terms: conditions — Irritable Bowel Syndrome; Negotiating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of the study is to investigate the clinical real-world effectiveness of a specific exposure based psychological treatment for irritable bowel syndrome (IBS). A secondary aim of the study is to find mediators of the treatment effect and thereby learn something about the working mechanism of the treatment.

DETAILED DESCRIPTION:
IBS is a debilitating disorder with a prevalence of 10% world wide. For patients with severe forms of IBS where medication and other interventions have failed it can be useful to try psychological treatment. National Institute for Health and Care Excellence (NICE) guidelines recommend cognitive behavior therapy or hypnotherapy.

Our research group at the Karolinska Institute in Stockholm has developed a cognitive behavioral treatment protocol for IBS. This treatment contains exposure therapy and mindfulness based exercises alongside psychoeducation. The treatment has been tested in four earlier randomized controlled trials (RCT) and produced large effect sizes compared to wait-list and moderate effect sizes compared to other active treatments or placebo.

The present study aims to examine the effectiveness of the treatment protocol under real-world circumstances at a secondary-care unit in Stockholm.

The Internet psychiatry Unit (IPSY) has been operative since 2007 and is run by Region Stockholm (i.e. the responsible authority for all publicly-funded healthcare in Stockholm). Patients with IBS have been treated at the clinic since 2015 and the treatment is delivered via an online treatment platform. The study is based on the clinics own data that has been collected for quality improvement reasons. Another aim of the study is to find out more about the working mechanisms behind the treatment by examining the weekly reports on behavioral avoidance and and anxiety that the patients file during treatment. All patients that have been treated at the clinic so far will be included in the study (N=319). Data has been collected between April 2015 and January 2022.

The study has an approved ethical permit from the Swedish Authority for Ethical Approvals.

The first hypothesis is that the treatment will be as effective in clinical routine care as it has been in earlier trials with a moderate to large effect-size from pre treatment to follow-up, six month after treatment. A second hypothesis is that the treatment effect is mediated by a change in behavioral avoidance that precedes symptomatic improvement.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IBS made by a licenced physician
* Able to provide written certificate of the diagnosis
* At least 16 years of age
* Daily access to computer, mobile phone or tablet with internet
* Account at health care guide 1177
* Proficient in Swedish

Exclusion Criteria:

* Considered having a high risk for suicide
* Unable to read or communicate in written form
* Do not understand Swedish language
* has planned to be away for more than 2 weeks during the treatment period
* suffers from another somatic or psychiatric condition needing to be prioritized or that might hinder treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that were treated for IBS at the Internet psychiatry unit in Stockholm from the opening of the unit (april 2015) until january 2022.
  The study population is believed to be representative of Swedish IBS-patients that have undergone the first steps of treatment for IBS (i.e. life style counseling, dietary advice and tried various medications) but still suffer significantly from their symptoms.
Sampling Method: Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
The Gastrointestinal Symptom Rating Scale for IBS (GSRS-IBS) | pre treatment (same day as treatment starts),
  It is a self-rating scale with 13 questions regarding the severity of the IBS-symptoms. The questions can be rated from 1-7, where 1 represents no discomfort at all and 7 means very severe discomfort. The total score may range from 13-91. The GSRS-IBS has demonstrated good psychometric properties for the different symptoms that are assessed, with an internal consistency (Cronbach's a) of .88 [17] and test-retest reliability between .55 and .70
Change from baseline IBS-symptoms measured with The Gastrointestinal Symptom Rating Scale for IBS (GSRS-IBS) | weekly during treatment (ten times in total, during the ten week long treatment)
  It is a self-rating scale with 13 questions regarding the severity of the IBS-symptoms. The questions can be rated from 1-7, where 1 represents no discomfort at all and 7 means very severe discomfort. The total score may range from 13-91. The GSRS-IBS has demonstrated good psychometric properties for the different symptoms that are assessed, with an internal consistency (Cronbach's a) of .88 [17] and test-retest reliability between .55 and .70
The Gastrointestinal Symptom Rating Scale for IBS (GSRS-IBS) | post treatment (same day as treatment ends). 10 weeks after treatment start.
  It is a self-rating scale with 13 questions regarding the severity of the IBS-symptoms. The questions can be rated from 1-7, where 1 represents no discomfort at all and 7 means very severe discomfort. The total score may range from 13-91. The GSRS-IBS has demonstrated good psychometric properties for the different symptoms that are assessed, with an internal consistency (Cronbach's a) of .88 [17] and test-retest reliability between .55 and .70
The Gastrointestinal Symptom Rating Scale for IBS (GSRS-IBS) | follow-up (six months after the treatment ended),
  It is a self-rating scale with 13 questions regarding the severity of the IBS-symptoms. The questions can be rated from 1-7, where 1 represents no discomfort at all and 7 means very severe discomfort. The total score may range from 13-91. The GSRS-IBS has demonstrated good psychometric properties for the different symptoms that are assessed, with an internal consistency (Cronbach's a) of .88 [17] and test-retest reliability between .55 and .70

SECONDARY OUTCOMES:
The Irritable bowel Syndrome - Behavioral Responses Questionnaire (IBS-BRQ) | pre treatment (same day as treatment starts)
  A scale measuring avoidance behavior and IBS-related anxiety'. The scale consists of 26 questions regarding food habits and toilet and social situations. The questions can be scored from 1-7 where 1 represents no control or avoidance behavior and 7 represents maximum avoidance or control, rendering a total score between 26 and 182. The IBS-BRQ has demonstrated excellent psychometric properties, with high internal consistency (Cronbach's alpha " .86) and high correlations with measures of dysfunctional IBS-related cognitions, IBS impact and impairment, anxiety, and depression
Change from baseline avoidance behaviors measured with The Irritable bowel Syndrome - Behavioral Responses Questionnaire (IBS-BRQ) | weekly during treatment (ten times in total, during the ten week long treatment)
  A scale measuring avoidance behavior and IBS-related anxiety'. The scale consists of 26 questions regarding food habits and toilet and social situations. The questions can be scored from 1-7 where 1 represents no control or avoidance behavior and 7 represents maximum avoidance or control, rendering a total score between 26 and 182. The IBS-BRQ has demonstrated excellent psychometric properties, with high internal consistency (Cronbach's alpha " .86) and high correlations with measures of dysfunctional IBS-related cognitions, IBS impact and impairment, anxiety, and depression
The Irritable bowel Syndrome - Behavioral Responses Questionnaire (IBS-BRQ) | post treatment (same day as treatment ends), ten weeks after treatment start
  A scale measuring avoidance behavior and IBS-related anxiety'. The scale consists of 26 questions regarding food habits and toilet and social situations. The questions can be scored from 1-7 where 1 represents no control or avoidance behavior and 7 represents maximum avoidance or control, rendering a total score between 26 and 182. The IBS-BRQ has demonstrated excellent psychometric properties, with high internal consistency (Cronbach's alpha " .86) and high correlations with measures of dysfunctional IBS-related cognitions, IBS impact and impairment, anxiety, and depression
The Irritable bowel Syndrome - Behavioral Responses Questionnaire (IBS-BRQ) | follow-up (six months after the treatment ended),
  A scale measuring avoidance behavior and IBS-related anxiety'. The scale consists of 26 questions regarding food habits and toilet and social situations. The questions can be scored from 1-7 where 1 represents no control or avoidance behavior and 7 represents maximum avoidance or control, rendering a total score between 26 and 182. The IBS-BRQ has demonstrated excellent psychometric properties, with high internal consistency (Cronbach's alpha " .86) and high correlations with measures of dysfunctional IBS-related cognitions, IBS impact and impairment, anxiety, and depression
Visceral Sensitivity Index (VSI) | pre treatment (same day as treatment starts)
  a scale designed to measure gastrointestinal specific anxiety (GSA; i.e., distress, avoidance, and safety behaviors in response to IBS-related stimuli). The VSI contains 15 items, which are scored between 0 and 5, rendering a total score between 0 (minimum GSA) and 75 (maximum GSA). The VSI has demonstrated high internal consistency (Cronbach's a = .90-.92) and has been shown to be associated with symptom severity and diagnostic status of IBS and also to be a mediator of the effect of exposure-based cognitive behavioral treatment on IBS symptoms
Visceral Sensitivity Index (VSI) | post treatment (same day as treatment ends), ten weeks after treatment start.
  a scale designed to measure gastrointestinal specific anxiety (GSA; i.e., distress, avoidance, and safety behaviors in response to IBS-related stimuli). The VSI contains 15 items, which are scored between 0 and 5, rendering a total score between 0 (minimum GSA) and 75 (maximum GSA). The VSI has demonstrated high internal consistency (Cronbach's a = .90-.92) and has been shown to be associated with symptom severity and diagnostic status of IBS and also to be a mediator of the effect of exposure-based cognitive behavioral treatment on IBS symptoms
Visceral Sensitivity Index (VSI) | follow-up (six months after the treatment ended)
  a scale designed to measure gastrointestinal specific anxiety (GSA; i.e., distress, avoidance, and safety behaviors in response to IBS-related stimuli). The VSI contains 15 items, which are scored between 0 and 5, rendering a total score between 0 (minimum GSA) and 75 (maximum GSA). The VSI has demonstrated high internal consistency (Cronbach's a = .90-.92) and has been shown to be associated with symptom severity and diagnostic status of IBS and also to be a mediator of the effect of exposure-based cognitive behavioral treatment on IBS symptoms
EuroQoL (EQ-5D) | pre treatment (same day as treatment starts)
  The EQ-5D consists of two parts: the health states descriptive system and the visual analog rating scale (VAS). In our study we used only the VAS scale which can be rated from 0-100. The endpoints of the VAS are labeled "best imaginable health state" and "worst imaginable health state" anchored at 100 and 0, respectively.
EuroQoL (EQ-5D) | post treatment (same day as treatment ends), ten weeks after treatment start.
  The EQ-5D consists of two parts: the health states descriptive system and the visual analog rating scale (VAS). In our study we used only the VAS scale which can be rated from 0-100. The endpoints of the VAS are labeled "best imaginable health state" and "worst imaginable health state" anchored at 100 and 0, respectively.
EuroQoL (EQ-5D) | follow-up (six months after the treatment ended)
  The EQ-5D consists of two parts: the health states descriptive system and the visual analog rating scale (VAS). In our study we used only the VAS scale which can be rated from 0-100. The endpoints of the VAS are labeled "best imaginable health state" and "worst imaginable health state" anchored at 100 and 0, respectively.
Short Form Health Survey (SF-12) | pre treatment (same day as treatment starts)
  This is a generic health status measure that includes both the physical domain and the mental domain of health. The scale has 12 items and has shown to be a reliable indicator of subjectively perceived health (Jenkinson C, et al., 1990).
Short Form Health Survey (SF-12) | post treatment (same day as treatment ends), ten weeks after treatment start.
  This is a generic health status measure that includes both the physical domain and the mental domain of health. The scale has 12 items and has shown to be a reliable indicator of subjectively perceived health (Jenkinson C, et al., 1990).
Change from baseline health status measured with Short Form Health Survey (SF-12) | weekly during treatment (ten times in total, during the ten week long treatment)
  This is a generic health status measure that includes both the physical domain and the mental domain of health. The scale has 12 items and has shown to be a reliable indicator of subjectively perceived health (Jenkinson C, et al., 1990).
Short Form Health Survey (SF-12) | follow-up (six months after the treatment ended)
  This is a generic health status measure that includes both the physical domain and the mental domain of health. The scale has 12 items and has shown to be a reliable indicator of subjectively perceived health (Jenkinson C, et al., 1990).

CONTACTS AND LOCATIONS:
Overall Officials: Brjánn Ljótsson, Ass. Prof., Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared due to General Data Protection Regulation (GDPR). Researchers that want to share the data must apply for ethical permit from The Authority for Ethical Approvals in Sweden.

REFERENCES:
- [Background] Jenkinson C, Layte R, Jenkinson D, Lawrence K, Petersen S, Paice C, Stradling J. A shorter form health survey: can the SF-12 replicate results from the SF-36 in longitudinal studies? J Public Health Med. 1997 Jun;19(2):179-86. doi: 10.1093/oxfordjournals.pubmed.a024606. PMID 9243433
- [Derived] Wallen H, Ljotsson B, Lindfors P, Forsell E, Hesser H, Svanborg C. Internet-Delivered Exposure-Based Cognitive Behavior Therapy for Irritable Bowel Syndrome: A Clinical Effectiveness Study. Am J Gastroenterol. 2025 Apr 1;120(4):856-863. doi: 10.14309/ajg.0000000000003059. Epub 2024 Aug 28. PMID 39194012